CLINICAL TRIAL: NCT01295398
Title: Influence of the Nebulizer on the Clinical Efficacy of Hypertonic Saline 3% in Children Aged Less Than 18 Months and Hospitalized With Acute Viral Bronchiolitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2010-A01237-32; 2010-24 (Other: AP HM)
Record Dates: First submitted 2011-02-09; First posted 2011-02-14 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2011-03

CONDITIONS: Acute Viral Bronchiolitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- conventional jet-nebulizer (Other): (particles diameter of 4-5 µm)
  Interventions: Device: nebulisations
- a jet-nebulizer adapted for infants (Experimental): (particles diameter of 2-2.5 µm),
  Interventions: Device: nebulisations
- a mesh-nebulizer adapted for infants (Experimental): (particles diameter of 2-2.5 µm).
  Interventions: Device: nebulisations

INTERVENTIONS:
Device: nebulisations

SUMMARY:
The aim of the investigators study is to compare in children aged less than 18 months and hospitalized for an acute viral bronchiolitis the efficacy of the HS 3% (Mucoclear®, sterile ampoules of 4 ml) nebulised with a conventional jet-nebulizer (particles diameter of 4-5 µm), or with a jet-nebulizer adapted for infants (particles diameter of 2-2.5 µm), or with a mesh-nebulizer adapted for infants (particles diameter of 2-2.5 µm).

ELIGIBILITY:
Inclusion Criteria:

* Infant of less than 18 months old
* infant hospitalized for a 1st episode of bronchiolitis defined as a 1st episode of respiratory difficulty with sibilant and\or crépitants in a viral context (head cold and\or cough and\or fever and\or notion of contage)
* Necessity of an clinical score upper to 4. This clinical score, described by Wang in 1992, is the clinical score classically used in the studies concerning the acute(sharp) bronchiolitis of the infant ( 8,9,12 ). He(it) is at most on 12 points.
* absence of respiratory décompensation requiring an admission in Unity of Pediatric Intensive care
* signature of the Informed consent
* Membership in a national insurance

Exclusion Criteria:

* Refusal of the parents to participate in the study
* 18-month-old infant hospitalized for acute(sharp) bronchiolitis with a clinical score lower than 4.
* signs of respiratory décompensation requiring a transfer in resuscitation, signs of hypercapnie or episodes of apneas
* histories of bronchiolitis or asthma of the infant
* cardiac underlying pathology, respiratory, neuromuscular, immunodeficient or former premature of less of 34 weeks of amenorrhoea and less than 3 months of corrected age.
* child having set within 6 hours preceding the inclusion a treatment by bronchodilatateurs or corticoids by systematic or inhaled way.

Ages: 28 Days to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 168 (Estimated)
Dates: Start 2010-12; Primary Completion 2014-05 (Actual); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
the improvement of the clinical score of severity at the 48th hour between the 3 groups of children | 12 months

SECONDARY OUTCOMES:
the number of children requiring oxygen | 12 months
tolerance of the nebulisations | 12 months
the number of complications. | 12 months
the number of parenteral nutrition | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: BERNARD BELAIGUES, Study Director — Assistance Publique hôpitaux de Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France